CLINICAL TRIAL: NCT00190086
Title: Syndrome X and Endothelial Dysfunction
Status: Terminated | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Other Study IDs: FEMH-94001
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2001-12

CONDITIONS: Syndrome X
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Cardiac syndrome X is characterized by angina, positve stress test, and patent coronary angiography, and its probable mechanism is microvascular dysfunction associated with endothelial dysfunction. We used brachial artery flow-mediated vasodilation to assess the endothelial function of the patients with syndrome X, coronary artery disease, and controls. Methods: We enrolled 28 patients with syndrome X, 11 healthy volunteers and 11 coronary artery disease patients. All subjects underwent a 2-step brachial artery flow-related vasodilation test: ultrasound artery diameter was measured at rest and after occlusion to assess endothelium-dependent vasodilation and after sublingual nitroglycerin to determine endothelium-independent condition. Serum endothelin-1 assay was performed for all participants. Results: The cardiac syndrome X patients had lower brachial artery dilation ratio (diameter after test/ diameter before test) than controls (1.10 +/- 0.09 versus 1.27 +/- 0.11, p=0.013), but the ratio is still higher than CAD patients (1.10 +/- 0.09 versus 1.02 +/- 0.07, p<0.001). After sublingual nitroglycerin, all 50 subjects had adequate vasodilation. Besides, normal controls have higher endothelin-1 level than the others.

We concluded that syndrome X patients have worse endothelial function than healthy control, but patients of CAD had even worse endothelium function than cardiac syndrome X patients.

Keywords: Cardiac syndrome X, coronary artery disease, endothelium-dependent vasodilation, endothelium-independent vasodilation, flow-mediated vasodilation, endothelin-1

DETAILED DESCRIPTION:
Cardiac syndrome x (CSX), which is defined as the combination of typical chest pain, electrocardiography or nuclear medicine evidence suggesting myocardial ischemia, and patent coronary arteriogram, comprises approximately 10-30% of the patients undergoing coronary angiogram.1,2 However, since it was first introduced in 1973, the pathogenesis of CSX has remained an enigma.1, 2 Among all the hypothetic explanations of CSX, including abnormal pain perception and non-cardiogenic origin of pain, the coronary microvascular dysfunction (microvascular angina), which represents reduced microvascular dilatory response and increased resistence, has been consistently found in CSX patients. 2, 3 This microvascular angina is believed to bridge the gap between the ischemic evidence and the normal-looking of coronary tree of CSX, and seems attributed to the endothelium dysfunction (ED), another frequently reported abnormality in CSX.2.3 By definition, ED is characterized by the endothelium-dependent vasodilation (EDVD) impairment, which is believed to be caused by decreased release of NO activity and/or activity, while the endotheliumindependent vasodilation (EIVD) remains preserved. 2,3,4 Therefore, it is asserted that endothelium-dependent dilatation of the resistance coronary arteries is defective in patients with CSX, and such defects may contribute to the altered regulation of myocardial perfusion in these patients.5 On the other hand, ED play a pivotal role in the development, progression, and clinical manifestations of atherosclerosis, as well as in the development of ischemia and thrombosis in the late stages of the disease, by promoting coronary vasoconstriction and thrombosis.4 Instead of using invasively intravascular measuring method used for endothelial function assessment, Celermajer et al first introduced the non-invasive measurement of the flow-mediated vasodilation (FMD) of forearm brachial artery in the assessment of EDVD and EIVD.6 This method was reported to have good correlation to the invasively intravascular studies in coronary systems.4 In this study, we want to compare the difference of forearm FMD, which respond to specially programmed stimuli, in three patient groups: CSX, coronary artery disease (CAD), and normal volunteers. A two-staged stimulation strategy is utilized to assess the EDVD (with cuff occlusion) and EIVD (with sublingual nitroglycerin) consecutively. A baseline plasma endothelin-1 (ET-1) concentration is also checked for each patient enrolled.

ELIGIBILITY:
Inclusion Criteria:

* which was performed under the impression of CAD due to positive treadmill electrocardiography test or ischemic evidence on Thallium scan, yielded the result of patent coronary tree. After the confirmation of angina symptoms and double-blinded review of the stress test and angiography result by 2 cardiologists to exclude controversial result

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28
Dates: Start 2001-01; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: A H Li, MD, Principal Investigator — Far Eastern Memorial Hospital